CLINICAL TRIAL: NCT00783302
Title: A Prospective, Multi-Center Registry Study for Clinical Outcome in Subjects Undergoing Coronary Computed Tomography Angiography (CCTA) Examination (VISIPAQUE Registry Study)
Brief Title: Study in Subjects Suspected of Having CAD Undergoing VISIPAQUE-enhanced CCTA as Part of Their Routine Medical Care
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: GE-012-096
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: CAD; Visipaque; CCTA
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess prognostic value of CCTA examination in subjects who undergo CCTA as part of their medical care when compared to a standard of truth, i.e. subject outcomes during each follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* The subject is over 18 years old, exhibits chest pain syndrome and is scheduled to undergo a VISIPAQUE-enhanced CCTA examination for one of the following reasons:- Intermediate pre-test probability of CAD.
* An uninterruptible/equivocal stress test (exercise, perfusion, or stress echo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient suspected of having coronary artery disease or CAD.
Sampling Method: Non-Probability Sample
Enrollment: 885 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Sheng, M.D., Principal Investigator — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 885 subjects enrolled in the Study. 874 subjects are in the safety population where adverse event data was collected, 857 subjects are in the efficacy population. 850 subjects completed the study. 35 subjects discontinued the study.
Groups:
- Arm 1: Visipaque Injection x 320mgI/mL: Injection of Visipaque at a concentration of 320mg I /mL.
Period: Overall Study
Arm/Group | Arm 1: Visipaque Injection x 320mgI/mL
Started | 885
Completed | 850
Not Completed | 35
Not completed — Lost to Follow-up | 17
Not completed — Technical Problems | 11
Not completed — Protocol Violation | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: Visipaque Injection x 320mgI/mL
Number analyzed (Participants) | 874
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.96)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 568
  >=65 years | 306
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 431
  Male | 443
Region of Enrollment [Number; unit: participants]
  United States | 736
  Canada | 138

OUTCOME MEASURES:

1. Primary Outcome: The Sensitivity of Visipaque-enhanced Coronary Computed Tomography Angiography (CCTA) for Predicting Downstream Cardiovascular Events at Each Follow-up Period When Compared to the Standard of Truth (SoT).
Description: Statistical analysis of the Sensitivity of Visipaque-enhanced CCTA for predicting downstream cardiovascular events at each follow-up period when compared to the SoT. The results are calculated as percentage of participants.
Time Frame: Within 1 month, 6 months and 12 months post contrast administration.
Population: The subject follow-up period went from 1 month, 6 months and 12 months.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Groups:
- Sensitivity - Subject Follow-up Period 1 Month; Sensitivity - Subject Follow-up Period 6 Months; Sensitivity - Subject Follow-up Period 12 Months: Number of Subjects Positive by Coronary Computed Tomography Angiography (CCTA) & Standard of Truth (SoT) / # Subjects Negative by Standard of Truth (SoT).
Arm/Group | Sensitivity - Subject Follow-up Period 1 Month | Sensitivity - Subject Follow-up Period 6 Months | Sensitivity - Subject Follow-up Period 12 Months
Number analyzed (Participants) | 51 | 71 | 76
Percentage of Subjects | 96.1 [86.5 to 99.5] | 95.8 [88.1 to 99.1] | 94.7 [87.1 to 98.5]

2. Primary Outcome: The Positive Predictive Value (PPV) of Visipaque-enhanced Coronary Computed Tomography Angiography (CCTA) for Ruling Out Downstream Cardiovascular Events at Each Follow-up Period When Compared to the Standard of Truth (SoT).
Description: Statistical analysis of the Positive Predictive Value (PPV) of Visipaque-enhanced CCTA for predicting downstream cardiovascular events at each follow-up period when compared to the SoT.The results are calculated as percentage of participants.
Time Frame: Within 1 month, 6 months and 12 months post contrast administration.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Groups:
- Positive Predictive Value - Subject Follow-up Period 1 Month; Positive Predictive Value - Subject Follow-up Period 6 Months; Positive Predictive Value - Subject Follow-up Period 12 Months: Number of Subjects True Positive by Coronary Computed Tomography Angiography (CCTA) / # Subjects Positive by Coronary Computed Tomography Angiography (CCTA)
Arm/Group | Positive Predictive Value - Subject Follow-up Period 1 Month | Positive Predictive Value - Subject Follow-up Period 6 Months | Positive Predictive Value - Subject Follow-up Period 12 Months
Number analyzed (Participants) | 174 | 173 | 172
Percentage of Subjects | 28.2 [21.6 to 35.5] | 39.3 [32.0 to 47.0] | 41.9 [34.4 to 49.6]

3. Primary Outcome: The Specificity of Visipaque-enhanced Coronary Computed Tomography Angiography (CCTA) for Ruling Out Downstream Cardiovascular Events at Each Follow-up Period When Compared to the Standard of Truth (SoT).
Description: Statistical analysis of the Specificity of Visipaque-enhanced CCTA for ruling out downstream cardiovascular events at each follow-up period when compared to the SoT.The results are calculated as percentage of participants.
Time Frame: Within 1 month, 6 months and 12 months post contrast administration.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Groups:
- Specificity - Subject Follow-up Period 1 Month; Specificity - Subject Follow-up Period 6 Months; Specificity - Subject Follow-up Period 12 Months: Number of Subjects Negative by Coronary Computed Tomography Angiography (CCTA) & Standard of Truth (SoT) / # Subjects Negative by Standard of Truth (SoT).
Arm/Group | Specificity - Subject Follow-up Period 1 Month | Specificity - Subject Follow-up Period 6 Months | Specificity - Subject Follow-up Period 12 Months
Number analyzed (Participants) | 806 | 782 | 767
Percentage of Subjects | 84.5 [81.8 to 86.9] | 86.6 [84.0 to 88.9] | 87.0 [84.4 to 89.3]

4. Primary Outcome: The Negative Predictive Value (NPV) of Visipaque-enhanced Coronary Computed Tomography Angiography (CCTA) for Ruling Out Downstream Cardiovascular Events at Each Follow-up Period When Compared to the Standard of Truth (SoT).
Description: Statistical analysis of the Negative Predictive Value (NPV) of Visipaque-enhanced CCTA for ruling out downstream cardiovascular events at each follow-up period when compared to the SoT.The results are calculated as percentage of participants.
Time Frame: Within 1 month, 6 months and 12 months post contrast administration.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Groups:
- Negative Predictive Value - Subject Follow-up Period 1 Month; Negative Predictive Value - Subject Follow-up Period 6 Months; Negative Predictive Value - Subject Follow-up Period 12 Months: Number of Subjects True Negative by Coronary Computed Tomography Angiography (CCTA) / # Subjects Negative by Coronary Computed Tomography Angiography (CCTA)
Arm/Group | Negative Predictive Value - Subject Follow-up Period 1 Month | Negative Predictive Value - Subject Follow-up Period 6 Months | Negative Predictive Value - Subject Follow-up Period 12 Months
Number analyzed (Participants) | 683 | 680 | 671
Percentage of Subjects | 99.7 [98.9 to 100.0] | 99.6 [98.7 to 99.9] | 99.4 [98.5 to 99.8]

5. Secondary Outcome: Summary of Subjects Developing 1 or More Positive and Negative Cardiac Clinical Outcomes at 1 Month, 6 Months, and 12 Months After Undergoing Coronary Computed Tomography Angiography (CCTA) Examination Using Visipaque.
Description: The number of subjects in the efficacy population developing 1 or more positive and negative cardiac clinical outcomes at 1 month, 6 months, and 12 months after undergoing a Coronary Computed Tomography Angiography (CCTA) examination using Visipaque. Clinical outcomes are independent of any serious adverse events and adverse events associated with the drug administration.
  This outcome measure is not reporting those subjects with serious adverse events and adverse events associated with the drug administration.
Time Frame: Within 1 month, 6 months and 12 months post contrast administration.
Measure: Number; unit: Number of Subjects
Groups:
- Follow-up Period at 1 Month: Summary of Patient-Level Clinical Outcomes by Follow-up Period (Efficacy Population) for 1 month.
- Follow-up Period at 6 Months: Summary of Patient-Level Clinical Outcomes by Follow-up Period (Efficacy Population) for 6 months.
- Follow-up Period at 12 Months: Summary of Patient-Level Clinical Outcomes by Follow-up Period (Efficacy Population) for 12 months.
Arm/Group | Follow-up Period at 1 Month | Follow-up Period at 6 Months | Follow-up Period at 12 Months
Number analyzed (Participants) | 857 | 853 | 843
Number of Subjects
  Positive Clinical Outcome | 51 | 71 | 76
  Negative Clinical Outcome | 806 | 782 | 767

ADVERSE EVENTS:
Description: Adverse event collection were taken from 874 subjects coming from the safety population of this study.
Arm/Group | Arm 1: Visipaque Injection x 320mgI/mL
Serious Adverse Events (participants affected / at risk) | 8/874
Other Adverse Events (participants affected / at risk) | 0/874
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Visipaque Injection x 320mgI/mL (N=874)
Angina Pectoris (Cardiac disorders) | 3 (3)
Coronary Artery Disease (Cardiac disorders) | 2 (2)
Coronary Artery Stenosis (Cardiac disorders) | 1 (2)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No